CLINICAL TRIAL: NCT00005946
Title: A Pilot Study of Combined Chemotherapy and Donor Lymphocyte Infusion for Hematologic Malignancies in Relapse After Allogeneic Bone Marrow Transplantation
Brief Title: Chemotherapy Plus Donor White Blood Cell Infusion in Treating Patients With Relapsed Hematologic Cancer Following Donor Peripheral Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: MSGCC-9951; CDR0000067863 (Registry Identifier: PDQ (Physician Data Query)); NCI-V00-1588
Record Dates: First submitted 2000-07-05; First posted 2004-03-05 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; recurrent/refractory childhood Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Filgrastim; Cyclophosphamide; Etoposide

INTERVENTIONS:
Biological: filgrastim
Biological: therapeutic allogeneic lymphocytes
Drug: cyclophosphamide
Drug: etoposide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. White blood cells from donors may be able to prevent graft-versus-host disease in patients with hematologic cancer that has relapsed following donor peripheral stem cell transplantation.

PURPOSE: Phase I trial to study the effectiveness of chemotherapy plus donor white blood cell infusion in treating patients who have relapsed hematologic cancer following donor peripheral stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the minimum amount of chemotherapy in combination with donor lymphocyte infusion required to obtain a rate of 30-60% graft versus host disease in patients with hematologic malignancies relapsed after allogeneic stem cell transplantation.

OUTLINE: This is a dose de-escalation study. Patients receive etoposide IV continuously on days 1-3; cyclophosphamide IV on day 8; donor lymphocyte infusion IV on day 10; and filgrastim (G-CSF) subcutaneously or IV beginning on day 10 and continuing until blood counts recover. Cohorts of 3-6 patients receive six de-escalating levels of chemotherapy until the minimum amount of chemotherapy in combination with donor lymphocyte infusion required to obtain a rate of 30-60% graft versus host disease (GVHD) is determined. The target dose level is defined as the level at which 2 of 6 patients develop GVHD, and the next lower dose level has no more than 1 patient experiencing GVHD. Patients are followed every 3 months for the first year, every 6 months for the second year, and yearly thereafter.

PROJECTED ACCRUAL: A total of 18-21 patients will be accrued over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed relapsed or refractory hematologic malignancy Acute leukemia Myelodysplasia Non-Hodgkin's lymphoma Hodgkin's disease Multiple myeloma Chronic lymphocytic leukemia Chronic myeloid leukemia Accelerated phase or blast crisis Chronic phase with failed prior donor lymphocyte infusion No active acute or extensive chronic graft versus host disease Prior allogeneic stem cell transplant (SCT) required At least 60 days since prior SCT Nonmyeloablative SCT allowed

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: Greater than 4 weeks Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No severe psychiatric illness that may preclude informed consent Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 7 days since prior immunomodulatory medications (e.g., interferon or interleukin-2) Chemotherapy: Not specified Endocrine therapy: At least 7 days since prior steroids Radiotherapy: Not specified Surgery: Not specified Other: At least 7 days since prior immunosuppressives (e.g., cyclosporine, tacrolimus, or mycophenolate mofetil) No concurrent immunosuppressive medications for graft versus host disease

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-10 (Actual); Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bijoyesh Mookerjee, MD, Study Chair — Jefferson Medical College of Thomas Jefferson University
Locations (1):
- Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland, United States